CLINICAL TRIAL: NCT04125069
Title: Role of Mitochondrial Dysfunction in the Occurrence of Acute Kidney Injury(AKI) in Postoperative Cardiac Surgery
Brief Title: Role of Mitochondrial Dysfunction in the Occurrence of Acute Kidney Injury (AKI) in Postoperative Cardiac Surgery
Acronym: MIT-CEC
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 18_RIPH3-24
Record Dates: First submitted 2019-10-09; First posted 2019-10-14 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Patients Undergoing Coronary Artery Bypass Graft (CABG) Surgery Requiring Extracorporeal Circulation
Keywords: Mitochondrial dysfunction; Acute Kidney Injury (AKI); Coronary Artery Bypass Graft (CABG) Surgery; Extracorporeal circulation; Inflammatory response; Type 2 diabete
MeSH Terms: conditions — Mitochondrial Diseases; Acute Kidney Injury | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged from 18 to 85 years: Cardiac surgery patients aged from 18 to 85 years,programmed for Coronary artery bypass graft requiring ECC.
  Interventions: Procedure: Coronary Artery Bypass Graft (CABG)

INTERVENTIONS:
Procedure: Coronary Artery Bypass Graft (CABG) — Mitochondrial function will be studied on cardiac tissue collected intraoperatively at the time of placement of the ECC cannulas by the surgeon. Fragments from auricle dissection of the right atrium of the patient will be requalified as sample residues, and will be used immediately by the surgeon to measure mitochondrial respiration (measurement of oxygen consumption by oxygenation and permeability test of the external mitochondrial membrane by the addition of cytochrome C in the oxygen chamber).

SUMMARY:
Cardiac Surgery and Acute Kidney Failure (AKI) post Surgery:

AKI is a frequent complication in the immediate aftermath of cardiac surgery with an incidence varying from 5 to 40%. KDIGO criteria (Kidney Disease: Improving Global Outcomes) are used to define the AKI in cardiac surgery because of their validated prognostic value in this patient population. The occurrence of a postoperative AKI, even of low severity, is accompanied by a significant increase in the duration of hospitalization and mortality. The AKI risk factors in cardiac surgery are related to the precarious clinical conditions of the patient before the surgery, to the complex surgical context, to the surgical procedures particularly the duration of extracorporeal circulation (ECC) greater than 120 min and the occurrence of a postoperative circulatory insufficiency.

AKI and inflammatory response:

The mechanisms involved in postoperative AKI in cardiac surgery, are low cardiac output, ischemia reperfusion injury (IRI), mechanical intravascular hemolysis, hypothermia, and activation of the neuroendocrine system by the ECC.

In addition, ECC triggers a secondary inflammatory response to blood contact with the ECC circuit and membranes. The secondary stimulation of immunocompetent cells accompanies secretion of many cytokines and proinflammatory mediators via the activation of nuclear transcription factors as the NFκB factor.

Of the 50 000 ECC performed per year in France, about 25% of the patients develop a Systemic Inflammatory Response Syndrome (SIRS). Although most often transient, SIRS can intensify and lead to a multi-visceral failure and to death, especially if the patient presents medical history of type 2 diabete. Increase of postoperative plasma cytokine levels has a positive predictive value on the occurrence of AKI and the risk of death.

Priming of the NLRP3 inflammasome and post ECC inflammatory response:

In addition to activation by nuclear transcription factors (NFκB), the inflammatory syndrome may develop secondarily to the activation of multi-protein platforms, called inflammasomes.

The activation of the NLRP3 inflammasome has been particularly studied in humans because of its association with multiple chronic inflammatory pathologies, infectious and cardio-metabolic diseases. Its activation is the combination of intracellular receptors like NOD-like receptors (NLR) types, ASC-like adapter proteins and pro caspase-1.

This assembly activates inflammatory caspases (caspase-1, in particular) responsible for the cleavage of pro-interleukins IL-1β and IL-18 in mature pro-inflammatory cytokines that participate in the orchestration of the inflammatory response.

Activation of the NLRP3 inflammasome requires prior priming which allows increase of NLRP3 and pro-cytokines IL1β and IL18 expressions. This priming is particularly intense in the presence of a mitochondrial dysfunction and of an increase in reactive oxygen species (ROS). Next, the activation of the NLRP3 inflammasome may be secondary to the presence of danger signals from cellular damages, such as cellular and mitochondrial debris (including mitochondrial DNA) recognized by NLRP3 receptors. Thus, preoperative mitochondrial dysfunction and its postoperative aggravation by ECC due to IRI induced by ECC represents powerful signals ,of the NLRP3 inflammasome activation.

Research hypothesis:

The hypothesis is that the preoperative priming of the NLRP3 inflammasome by a preoperative mitochondrial dysfunction is a factor favoring the occurrence of postoperative AKI after cardiac surgery with ECC.

For type 2 diabetic patients, the investigators think that preoperative mitochondrial dysfunction (mitochondrial respiration abnormalities and hyperpermeability of mitochondrial membranes) is accentuated worsening IRI induced by the ECC.

This increases postoperative release of cells and mitochondrial debris that maintain the activation of the NLRP3 inflammasome, exacerbating the inflammatory response and favoring the occurrence of AKI.

DETAILED DESCRIPTION:
Primary objective of the research:

Describe the association between preoperatives mitochondrial dysfunction markers and the occurrence of AKI in postoperative cardiac surgery with ECC.

Secondary objective of research:

Describe, in preoperative cardiac surgery, the level of mitochondrial dysfunction according to type 2 diabetic status (inflammation-promoting factor).

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 85 years old,
* Patients undergoing coronary artery bypass graft requiring circulation extracorporeal,
* Have been informed of the research,
* Having defended its decision of non-opposition to the research on samples taken during the treatment and on the data medical file,
* Patients affiliated to a social security scheme.

Exclusion Criteria:

* Pregnant or nursing woman,
* Diabetic type 1,
* Emergency cardiac surgery,
* Valvular replacement surgery,
* Clinical heart failure or ejection fraction of the ventricle left EFVG <50%,
* Valvular pathology,
* Left atrial dilation> 40 mm,
* Systolic pulmonary arterial pressure> 40 mmHg,
* BNP (Brain natriuretic peptide) level> 100 ng / L,
* Atrial fibrillation or flutter,
* Right coronary stenosis> 50%,
* Chronic renal failure defined by a filtration rate Glomerular GFR (GFR) less than 60 ml / min / 1.73 m2 estimated from creatinine by the equation CKD-EPI (Chronic Kidney Disease - Epidemiology Collaboration).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing coronary artery bypass graft requiring circulation extracorporeal
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Describe the correlation between preoperatives mitochondrial dysfunction markers and the occurrence of AKI in postoperative cardiac surgery with ECC. | 15 months
  Frequency of postoperative onset of an AKI defined according to KDIGO criteria according to preoperative mitochondrial dysfunction (preoperative levels of oxygen consumption by the mitochondria and permeability of the external mitochondrial membrane at Cytochrome CytC in heart tissue.
  KDIGO criteria will be used for diagnosis of AKI, defined as an increase in plasma creatinine ≥0.3 mg/dl (≥26.5 μmol/l) in the 48hours (or an increase of more than 1.5 to 1.9 times the baseline) and urine output <0.5 ml/kg/h in the last 6 to 12 hours.
Describe the correlation between preoperatives mitochondrial dysfunction markers and the occurrence of AKI in postoperative cardiac surgery with ECC. | 15 months
  To measure the mitochondrial respiration and to perform the permeability test of the mitochondrial external membrane, a high resolution oxygraph that can detect levels of mitochondrial respiration on few milligrams samples will be used (O2k, Oroboros, Innsbruck, Austria). Oxygen consumption fluxes will be expressed in pmol O2*s-1*mg-1 of dry tissue.

SECONDARY OUTCOMES:
Describe, in preoperative cardiac surgery, the level of mitochondrial dysfunction according to type 2 diabetic status (inflammation-promoting factor). | 15 months
  Diabetes will be diagnosed if the fasting blood glucose (8 hours) is equal to or greater than 1.26 g/l (7.0 mmol/l) twice or equal to or greater than 2 g/l at any time of the day.
  A measurement of glycated hemoglobin (HbA1c) will help to know the glycemic balance of two to three months before the patient inclusion. Diabetes will be considered balanced if the HbA1c level is between 6 and 8%.
Describe, in preoperative cardiac surgery, the level of mitochondrial dysfunction according to type 2 diabetic status (inflammation-promoting factor). | 15 months
  To measure the mitochondrial respiration and to perform the permeability test of the mitochondrial external membrane, a high resolution oxygraph that can detect levels of mitochondrial respiration on few milligrams samples will be used (O2k, Oroboros, Innsbruck, Austria). Oxygen consumption fluxes will be expressed in pmol O2*s-1*mg-1 of dry tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Rémi NEVIERE, PhD, Study Director — CHU de Martinique
Locations (1):
- CHU de Martinique, Fort-de-France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zakkar M, Ascione R, James AF, Angelini GD, Suleiman MS. Inflammation, oxidative stress and postoperative atrial fibrillation in cardiac surgery. Pharmacol Ther. 2015 Oct;154:13-20. doi: 10.1016/j.pharmthera.2015.06.009. Epub 2015 Jun 24. PMID 26116810
- [Background] Corral-Velez V, Lopez-Delgado JC, Betancur-Zambrano NL, Lopez-Sune N, Rojas-Lora M, Torrado H, Ballus J. The inflammatory response in cardiac surgery: an overview of the pathophysiology and clinical implications. Inflamm Allergy Drug Targets. 2015;13(6):367-70. doi: 10.2174/1871528114666150529120801. PMID 26021321
- [Background] Hoste EAJ, Vandenberghe W. Epidemiology of cardiac surgery-associated acute kidney injury. Best Pract Res Clin Anaesthesiol. 2017 Sep;31(3):299-303. doi: 10.1016/j.bpa.2017.11.001. Epub 2017 Nov 8. PMID 29248137
- [Background] Wang Y, Bellomo R. Cardiac surgery-associated acute kidney injury: risk factors, pathophysiology and treatment. Nat Rev Nephrol. 2017 Nov;13(11):697-711. doi: 10.1038/nrneph.2017.119. Epub 2017 Sep 4. PMID 28869251
- [Background] Patel SS, Palant CE, Mahajan V, Chawla LS. Sequelae of AKI. Best Pract Res Clin Anaesthesiol. 2017 Sep;31(3):415-425. doi: 10.1016/j.bpa.2017.08.004. Epub 2017 Sep 6. PMID 29248147
- [Background] O'Neal JB, Shaw AD, Billings FT 4th. Acute kidney injury following cardiac surgery: current understanding and future directions. Crit Care. 2016 Jul 4;20(1):187. doi: 10.1186/s13054-016-1352-z. PMID 27373799
- [Background] Ortega-Loubon C, Fernandez-Molina M, Carrascal-Hinojal Y, Fulquet-Carreras E. Cardiac surgery-associated acute kidney injury. Ann Card Anaesth. 2016 Oct-Dec;19(4):687-698. doi: 10.4103/0971-9784.191578. PMID 27716701
- [Background] Rheinheimer J, de Souza BM, Cardoso NS, Bauer AC, Crispim D. Current role of the NLRP3 inflammasome on obesity and insulin resistance: A systematic review. Metabolism. 2017 Sep;74:1-9. doi: 10.1016/j.metabol.2017.06.002. Epub 2017 Jun 11. PMID 28764843
- [Background] Prochnicki T, Latz E. Inflammasomes on the Crossroads of Innate Immune Recognition and Metabolic Control. Cell Metab. 2017 Jul 5;26(1):71-93. doi: 10.1016/j.cmet.2017.06.018. PMID 28683296
- [Background] Feldman N, Rotter-Maskowitz A, Okun E. DAMPs as mediators of sterile inflammation in aging-related pathologies. Ageing Res Rev. 2015 Nov;24(Pt A):29-39. doi: 10.1016/j.arr.2015.01.003. Epub 2015 Jan 29. PMID 25641058
- [Background] Traba J, Sack MN. The role of caloric load and mitochondrial homeostasis in the regulation of the NLRP3 inflammasome. Cell Mol Life Sci. 2017 May;74(10):1777-1791. doi: 10.1007/s00018-016-2431-7. Epub 2016 Dec 10. PMID 27942750